CLINICAL TRIAL: NCT04971408
Title: Passive Heating as an Accessible and Tolerable Strategy to Improve the Inflammatory Profile and Cardiometabolic Health in People With Spinal Cord Injury
Brief Title: Impact of Passive Heat on Metabolic, Inflammatory and Vascular Health in Persons With Spinal Cord Injury
Acronym: SCIPHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B3724-P
Record Dates: First submitted 2021-07-09; First posted 2021-07-21 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injury; Chronic Inflammation; Glucose Metabolism; Endothelial Function
Keywords: spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: passive heat stress with water perfused heat suits and electrical heating blankets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Other): passive heat stress x1 visit then no intervention for 8 weeks. participants continue regular exercise habits as usual.
  Interventions: Other: control
- Passive heat stress (Experimental): After arm 1, passive heat stress 3x/week x8 weeks.
  Interventions: Other: passive heat stress

INTERVENTIONS:
Other: passive heat stress — as above
  Other Names: water perfused suit and electrical heating blanket
  Arms: Passive heat stress
Other: control — participant engage in activity as usual
  Arms: control

SUMMARY:
SCI results in higher incidence of heart disease and diabetes and heart disease is the most common cause of death. Chronic inflammation, deleterious changes in vascular structure and impaired glucose metabolism are risk factors that contribute to both heart disease and diabetes. While exercise can help reduce these risk factors, paralysis and impaired accessibility often precludes exercise in persons with SCI. New research in able-bodied persons demonstrates passive heating decreases inflammation and improves vascular function. Similar studies in persons with SCI suggest they may also have the same health benefits however these studies only investigated the impact of short term (one episode) passive heating (as opposed to repeated bouts). Repeated bouts of heat exposure will likely be required to impact chronic inflammation, but this has never been tested in persons with SCI. This study will test the impact of repeated bouts (3x/week) of passive heat stress over a longer term (8 weeks) on inflammation, metabolism and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Stable SCI over 1 year of duration

Exclusion Criteria:

* Persons who smoke cigarettes
* Daily administration of anti-inflammatory medications
* Daily administration of vasoactive medications
* Pressure ulcer stage 3 or 4
* History of heat related illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
inflammatory markers | change from 0 to 8 to 16 weeks
  IL-6

SECONDARY OUTCOMES:
endothelial function | change from 0 to 8 to 16 weeks
  cutaneous vascular conductance measured via laser doppler flowmetry
glucose metabolism via oral glucose tolerance test | change from 0 to 8 to 16 weeks
  oral glucose tolerance test
inflammatory marker | change from 0 to 8 to 16 weeks
  TNF-alpha
inflammation | change from 0 to 8 to 16 weeks
  IL-1 beta
inflammation | change from 0 to 8 to 16 weeks
  IL-10
inflammation | change from 0 to 8 to 16 weeks
  Heat shock protein 72

OTHER OUTCOMES:
Health Related Quality of Life | change from 0 to 8 to 16 weeks
  RAND -36 survey
Chronic pain | change from 0 to 8 to 16 weeks
  SCI Pain Questionnaire
Mental Health | change from 0 to 8 to 16 weeks
  Mental Health Inventory-5

CONTACTS AND LOCATIONS:
Overall Officials: Michelle B Trbovich, MD, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (1):
- South Texas Health Care System, San Antonio, TX, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04971408/ICF_000.pdf